CLINICAL TRIAL: NCT03086759
Title: Intra-Articular Use of Platelet Rich Plasma Versus Corticosteroid: A Clinical Trials in Osteoarthritis of Knee.
Brief Title: Intra-Articular Platelet Rich Plasm Use in Osteoarthritis of Knee.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Nunes Tamashiro, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP UNIFESP 842 167/2014
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — triamcinolone hexacetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelet rich plasm group (Experimental)
  Interventions: Procedure: platelet rich plasm
- Triamcinolone Hexacetonide group (Active Comparator)
  Interventions: Drug: Triamcinolone Hexacetonide
- Isotonic Saline Solution group (Placebo Comparator)
  Interventions: Procedure: Isotonic Saline Solution

INTERVENTIONS:
Procedure: platelet rich plasm — intra-articular infiltration with platelet rich plasm
  Arms: Platelet rich plasm group
Drug: Triamcinolone Hexacetonide — intra-articular infiltration withTriamcinolone Hexacetonide
  Arms: Triamcinolone Hexacetonide group
Procedure: Isotonic Saline Solution — intra-articular infiltration with Isotonic Saline Solution
  Arms: Isotonic Saline Solution group

SUMMARY:
Osteoarthritis of the knee is a very prevalent disease. However, there are few therapeutic options for its patients. Platelet-rich plasma is a treatment option for chronic pain. If proven to be effective in its intra-articular use, Platelet-rich plasma may help in the treatment of these patients.

Goal:

Primary objective: To compare effectiveness in improving pain and function and the medium-term tolerance (12 weeks) of intra-articular injection of Platelet-rich plasma versus intraarticular injection of triamcinolone hexacetonide in patients with symptomatic primary knee osteoarthritis.

Secondary objective: To compare the medium-term effectiveness of intra-articular injection of Platelet-rich plasma versus intra-articular injection of triamcinolone hexacetonide to improve synovial hypertrophy and quality of life in these patients.

Methods: A prospective randomized controlled double-blind study with three groups (each with n = 33) of patients with symptomatic osteoarthritis of knees who will receive intra-articular infiltration in a single moment. Patients will be allocated to one of three groups: 1) Platelet-rich plasma group: patients who will receive plasma; 2) triamcinolone hexacetonide Group: patients who will receive 40mg of triamcinolone hexacetonide; And 3) Isotonic saline solution group: patients who will receive isotonic saline solution. The patients will be evaluated by "blind" evaluators in 4 assessment times up to 12 weeks of follow-up through clinical assessment instruments (rest and movement pain, joint edema, goniometry, clinical improvement scale, quality of life questionnaire as the SF36), functional (Womac questionnaire, M. Lequesne Functional Knee Index, 6 min walk test, Time up and go test), and ultrasound test (quantitative and semiquantitative measurement of synovial hypertrophy and semiquantitative Power Doppler).

Statistics: The following statistical tests will be used according to the need: Student's t test, Mann-whitney, Pearson's chi-square test and ANOVA for repeated measures. A statistical significance of 5% will be considered.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis
* degree II and II in Kellgren & Lawrence classification
* pain duration: more than three months
* pain in the visual analogue scale between 4 and 8cm
* agree in participate and sign the consent form

Exclusion Criteria:

* secondary knee osteoarthritis
* skin lesion in knee
* intraarticular joint injection in the previous three months
* steroids use in the previous 30 days
* degree I or IV in Kellgren & Lawrence classification
* inflammatory arthritis, gout and pseudo-gout
* cancer
* previous surgery in knee
* cardiovascular and respiratory disease that change functional status
* pregnancy and breastfeed
* coagulation disturb
* bacterial infection
* handicapped
* NSAIDs and Platelet anticoagulant in the previous month

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
Change in pain | Baseline, after 4, 8, 12 and 48 weeks
  Evaluated using a visual analogue scale

SECONDARY OUTCOMES:
Change in joint edema | Baseline, after 4, 8, 12 and 48 weeks
  Evaluated using a visual analogue scale
Change in range of motion | Baseline, after 4, 8, 12 and 48 weeks
  Evaluated using goniometry
Change in a clinical improvement scale | Baseline, after 4, 8, 12 and 48 weeks
  Evaluated using an improvement scale
Change in quality of life | Baseline, after 4, 8, 12 and 48 weeks
  Using the SF-36 questionnaire
Change in functional capacity | Baseline, after 4, 8, 12 and 48 weeks
  Using the WOMAC questionnaire
Change in functional capacity | Baseline, after 4, 8, 12 and 56 weeks
  Using the M Lequesne questionnaire
Change in functional capacity | Baseline, after 4, 8, 12 and 48 weeks
  Using the six minute walk test
Change in functional capacity | Baseline, after 4, 8, 12 and 48 weeks
  Using the time to up and go test
Changing in quantitative and semiquantitative measurement of synovial hypertrophy and semiquantitative Power Doppler | Baseline, after 4, 8, 12 and 48 weeks
  Using an ultrasound exam

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil